CLINICAL TRIAL: NCT00037401
Title: Postprandial Lipemia and Endothelial Function in ACCORD- Ancillary to ACCORD
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1168; R01HL069190 (NIH)
Record Dates: First submitted 2002-05-16; First posted 2002-05-17 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2008-01

CONDITIONS: Atherosclerosis; Cardiovascular Diseases; Hypercholesterolemia; Heart Diseases
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases; Hypercholesterolemia; Heart Diseases

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
To compare the effects of statin therapy alone with statin plus fibrate therapy on several emerging risk factors for atherosclerotic cardiovascular disease in a representative subgroup of the ACCORD cohort that is being followed for cardiovascular endpoints.

DETAILED DESCRIPTION:
BACKGROUND:

The National Heart, Lung, and Blood Institute-supported ACCORD trial uses two connected 2x2 designs to test the efficacy of (a) optimal glucose control (HbA1c = 6.0%) versus standard control (HbA1c + 7.5%) in 10,000 patients with type 2 diabetes mellitus, (b) more intense systolic blood pressure control (120 mm Hg) versus less intense control (140 mm Hg) in 4,200 of those patients, and (c) combined low density lipoprotein cholesterol lowering, triglyceride lowering, and high density lipoprotein cholesterol raising versus only low density lipoprotein cholesterol lowering in 5,800 of those patients. The primary outcome for the overall ACCORD trial is a combination of non-fatal myocardial infarction, non-fatal stroke, and cardiovascular death. The comparison of lipid-altering therapies is carried out in the Lipid Arm of ACCORD, in which the 5,800 subjects are treated with simvastatin and, in addition, are randomly assigned to receive either fenofibrate or placebo. The main ACCORD trial measures only fasting blood samples for lipids, lipoprotein fractions, and apolipoproteins. The ancillary study compares the effects of simvastatin plus fenofibrate with the effects of simvastatin alone on postprandial lipemia in 250 ACCORD patients at 4 sites in the Northeast Network.

The study is in response to an initiative on Ancillary Studies in Heart, Lung, and Blood Disease Trials released in June, 2000.

DESIGN NARRATIVE:

The ancillary study compares the effects of simvastatin plus fenofibrate with the effects of simvastatin alone on postprandial lipemia in 250 ACCORD patients at 4 sites in the Northeast Network. In addition, the study compare the effects of the two treatment strategies on baseline and postprandial endothelial function, and on markers of coagulation, endothelial function, and oxidative stress. The ancillary study provides a unique opportunity to determine possible mechanisms whereby simvastatin plus fenofibrate therapy may be associated with reduced cardiovascular events in the overall ACCORD trial. The study is divided into three specific aims. Specific Aim A: To carry out high fat load studies of postprandial lipemia in patients who are participating in the Lipid Arm of the ACCORD trial and compare postprandial excursions of triglycerides, triglyceride-rich lipoproteins, retinyl palmitate, and remnant lipoprotein cholesterol in patients receiving fenofibrate plus simvastatin with those postprandial excursions in patients receiving only simvastatin. Specific Aim B: To determine brachial artery dilatation in response to increased blood flow post- forearm ischemia just prior to, and five hours after, ingestion of a high fat load in the two patient groups.and Specific Aim C: To determine baseline levels of PAI-1, fibrinogen and factor VII, and postprandial excursions of factor VII, sVCAM-1, sICAM-1, and sE-selectin in the two patient groups.

ELIGIBILITY:
No eligibility criteria

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-09; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry Ginsberg — Columbia University Health Sciences